CLINICAL TRIAL: NCT03806127
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Vibegron Administered Orally for 12 Weeks to Women With Irritable Bowel Syndrome
Brief Title: Study to Evaluate the Efficacy and Safety of Vibegron Administered Orally for 12 Weeks to Women With Irritable Bowel Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Urovant Sciences GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: URO-901-2001
Record Dates: First submitted 2019-01-14; First posted 2019-01-16 (Actual); Results first posted 2021-07-30 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; Irritable Bowel Syndrome with predominantly diarrhea (IBS-D); Irritable Bowel Syndrome with mixed episodes of diarrhea and constipation (IBS-M); Vibegron; Beta-3 adrenergic receptor (β3-AR); Pain
MeSH Terms: conditions — Irritable Bowel Syndrome; Constipation; Pain | interventions — N-(4-((5-(hydroxy(phenyl)methyl)pyrrolidin-2-yl)methyl)phenyl)-4-oxo-4,6,7,8-tetrahydropyrrolo(1,2-a)pyrimidine-6-carboxamide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vibegron 75 mg (Experimental): Participants will receive vibegron 75 milligrams (mg) orally once daily for 12 weeks.
  Interventions: Drug: Vibegron
- Placebo (Placebo Comparator): Participants will receive matching placebo orally once daily for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vibegron — oral administration
  Other Names: RVT-901; MK-4618; KRP-114V; URO-901
  Arms: Vibegron 75 mg
Drug: Placebo — oral administration
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy and safety of vibegron, a beta-3 adrenergic receptor (β3-AR) agonist, in the treatment of pain associated with irritable bowel syndrome (IBS) due to IBS with predominant diarrhea (IBS-D) or mixed episodes of diarrhea and constipation (IBS-M).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of irritable bowel syndrome (IBS) with predominantly diarrhea (IBS-D) or IBS with mixed episodes of diarrhea and constipation (IBS-M) according to the Rome IV criteria
* Has completed a colonoscopy according to the American Gastroenterological Association criteria, with no clinically significant findings in the last 5 years
* Has no clinically significant findings on a physical examination or clinical laboratory tests that could interfere with study participation or confound study assessments, in the opinion of the Investigator. Serum tissue transglutaminase antibody (IgA) must be negative. Fecal calprotectin testing is optional and should only be considered if there is a strong suspicion that the participant has inflammatory bowel disease (IBD) (eg, family history in a 1st degree relative, other genetic factors, etc.) or other organic disease, according to the clinical judgement of the investigator.

Exclusion Criteria:

* Diagnosis of IBS-C or IBS-U per Rome IV criteria
* History of chronic idiopathic constipation or functional constipation
* Structural abnormality of the gastrointestinal tract or a disease (e.g., known small intestine bacterial overgrowth) or condition that can affect gastrointestinal motility
* History of a gastrointestinal motility disorder other than IBS (e.g., gastroparesis, intestinal pseudo-obstruction, achalasia, Parkinsons disease, multiple sclerosis, spinal cord injury)
* Prior history of a gastrointestinal malignancy, inflammatory bowel disease, celiac disease
* Planned gastrointestinal or abdominal surgery within the next 6 months
* Co-existing gastroesophageal reflux disease or functional dyspepsia with symptoms predominant to IBS symptoms
* Symptoms or diagnosis of a medical condition other than IBS that may contribute to abdominal pain (e.g., interstitial cystitis; fibromyalgia currently being treated with pregabalin or gabapentin; and endometriosis with uncontrolled abdominal pain)

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2018-12-31 (Actual); Primary Completion 2020-09-25 (Actual); Study Completion 2020-10-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (41):
- United States (41):
  - Synexus Clinical Research US, Inc.-Simon Williamson Clinic, Birmingham, Alabama
  - Clinical Research Associates, Huntsville, Alabama
  - Alabama Medical Group, PC, Mobile, Alabama
  - Hope Research Institute, Chandler, Arizona
  - Synexus Clinical Research US, Inc. - East Valley Family Physicians, PLC, Chandler, Arizona
  - Synexus Clinical Research US, Inc. - Central Arizona Medical Associates, PC, Mesa, Arizona
  - Synexus Clinical Research US, Inc. - Desert Clinical Research, LLC, Mesa, Arizona
  - Synexus - Clinical Research Advantage, Inc. - Central Phoenix Medical Clinic LLC, Phoenix, Arizona
  - GW Research Inc - ClinEdge-PPDS, Chula Vista, California
  - Triwest Research Associates, LLC, La Mesa, California
  - VA Long Beach Healthcare System - NAVREF, Long Beach, California
  - Southern California Research Institute Medical Group, Inc., Los Angeles, California
  - Desta Digestive Disease Medical Center, San Diego, California
  - Medical Associates Research Group, Inc., San Diego, California
  - Torrance Clinical Research, Torrance, California
  - Medical Research Center of Connecticut LLC, Hamden, Connecticut
  - Mayo Clinic - Division of Gastroenterology, Jacksonville, Florida
  - Florida Center For Gastroenterology, Largo, Florida
  - Clinical Research Center of Florida, Pompano Beach, Florida
  - Palm Beach Research - ClinEdge - PPDS, West Palm Beach, Florida
  - RNA America, LLC, Sugar Hill, Georgia
  - Investigators Research Group, LLC, Indianapolis, Indiana
  - Mandeville Private Physician Group, LLC, Mandeville, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Clinical Research Institute of Michigan, Chesterfield, Michigan
  - Synexus Clinical Research US, Inc. - Rita B. Chuang, MD, LLC, Henderson, Nevada
  - Advanced Research Institute, Reno, Nevada
  - Atrium Healthcare Center for Digestive Health, Charlotte, North Carolina
  - Carolina Digestive Diseases, Greenville, North Carolina
  - East Carolina Gastroenterology, Jacksonville, North Carolina
  - Dayton Gastroenterology, Inc., Beavercreek, Ohio
  - Central Sooner Research, Norman, Oklahoma
  - Synexus Clinical Research US, Inc. - Anderson, Anderson, South Carolina
  - Chattanooga Medical Research Inc, Chattanooga, Tennessee
  - Clinical Research Solutions PC, Jackson, Tennessee
  - DHAT Research Institute, Garland, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Synexus Clinical Research US, Inc.-Plano, Plano, Texas
  - Synexus Clinical Research US, Inc. - Wasatch Peak Family Practice, Layton, Utah
  - Advanced Research Institute, South Ogden, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 806 participants screened for this study, 222 were randomized (after a 2-week, single-blind placebo Run-in Period), and 222 received 1 dose of double-blind study drug in the Treatment Period (Safety Set: placebo, N = 111; vibegron, N = 111).
Groups:
- Placebo: Participants received matching placebo, orally, once daily for 12 weeks. Participants were stratified by Baseline abdominal pain intensity (API) score (< 6 versus ≥ 6 on a 0- to 10-point numeric rating scale) and irritable bowel syndrome (IBS) subtype (IBS with predominant diarrhea [IBS-D] versus IBS with mixed episodes of diarrhea and constipation [IBS-M]).
- Vibegron 75 mg: Participants received vibegron 75 milligrams (mg), orally, once daily for 12 weeks. Participants were stratified by Baseline API score (< 6 versus ≥ 6 on a 0- to 10-point numeric rating scale) and IBS subtype (IBS-D versus IBS-M).
Period: Overall Study
Arm/Group | Placebo | Vibegron 75 mg
Started | 111 | 111
Completed | 90 | 99
Not Completed | 21 | 12
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Protocol Violation | 3 | 1
Not completed — Adverse Event | 3 | 0
Not completed — Unable to Complete Procedures | 0 | 1
Not completed — Pregnancy | 0 | 1
Not completed — Lost to Follow-up | 5 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Could Not Come Due to Covid | 1 | 0
Not completed — Prescribed Exclusionary Medication (Med) | 1 | 0
Not completed — Ran Out of Study Meds (Covid Quarantine) | 1 | 0
Not completed — Covid 19 Restrictions | 2 | 0
Not completed — Withdrawn Due to Work/School Schedule | 0 | 1
Not completed — Covid 19 Concern; Possible Site Closure | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline data are reported for all randomized participants who took at least one dose of double-blind study medication and had at least one evaluable post-randomization weekly abdominal pain intensity (API) score (i.e., where evaluable was considered a minimum of 5 diary entries in a week).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Vibegron 75 mg | Total
Number analyzed (Participants) | 108 | 111 | 219
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.6 (13.10) | 40.5 (13.88) | 40.1 (13.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 111 | 219
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 82 | 80 | 162
  Black or African American | 24 | 25 | 49
  Captured as Other | 1 | 3 | 4
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
Abdominal Pain Intensity Score (Stratified Strata) [Count of Participants; unit: Participants] — Stratified strata was based on the randomization stratifications. Participants were asked to rate their IBS-related abdominal pain at its worst in the past 24 hours on a 0- to 10-point numeric rating scale, where 0 = no pain and 10 = the worst possible pain.
  Participants
    < 6 | 77 | 78 | 155
    ≥ 6 | 31 | 33 | 64
IBS Subtype (Stratified Strata) [Count of Participants; unit: Participants] — Stratified strata was based on the randomization stratifications. The Rome IV criteria classifies IBS into 4 distinct subtypes based on predominant stool consistency: IBS with predominantly constipation (IBS-C), IBS with predominantly diarrhea (IBS-D), IBS with mixed episodes of diarrhea and constipation (IBS-M), and IBS with unknown subtype (IBS-U). IBS-D: ≥ 25% diarrhea and < 25% constipation. IBS-M: ≥ 25% constipation and ≥ 25% diarrhea.
  Participants
    IBS-D | 63 | 66 | 129
    IBS-M | 45 | 45 | 90

OUTCOME MEASURES:

1. Primary Outcome: Number of Irritable Bowel Syndrome (IBS) With Predominantly Diarrhea (IBS-D) Participants Who Were Abdominal Pain Intensity (API) Weekly Responders at Week 12
Description: An API Weekly Responder was defined as a participant who experienced a decrease in the weekly average of "worst abdominal pain in the past 24 hours" scores of at least 30% compared with the Baseline weekly average. A participant was considered a responder over Weeks 1 to 12 if they met the criteria for at least 50% of the weeks assessed (i.e., ≥6 weeks).
Time Frame: Baseline; Week 12
Population: Full Analysis Set for IBS-D participants: all randomized participants with IBS-D who who took at least one dose of double-blind study medication and had at least one evaluable post-randomization weekly API score (i.e., where evaluable was considered a minimum of 5 diary entries in a week)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Vibegron 75 mg
Number analyzed (Participants) | 63 | 66
Participants | 27 | 27
Statistical Analysis 1: Comparison: Placebo vs Vibegron 75 mg; Test type: Other; Cochran-Mantel-Haenszel (CMH) Difference = -1.9, 90% CI 2-sided [-16.1 to 12.3] — Difference in proportion and corresponding confidence interval were calculated using the CMH risk difference estimate stratified by randomized Baseline abdominal pain (< 6 versus ≥ 6) strata, with weights proposed by Greenland and Robins

2. Secondary Outcome: Number of Global Improvement Scale (GIS) Responders at Week 12 for All IBS Participants, Including IBS-D and IBS-M Participants
Description: Global improvement assessment asks participants to evaluate their current IBS status by asking the following question: How would you rate your IBS signs or symptoms overall over the past 7 days?: (1) significantly relieved; (2) moderately relieved; (3) slightly relieved; (4) unchanged; (5) slightly worse; (6) moderately worse; (7) significantly worse. A responder was defined as a participant who answered that their symptoms were either moderately relieved or significantly relieved. A participant with a missing GIS response was considered to be a non-responder.
Time Frame: Week 12
Population: Full Analysis Set: all randomized participants who took at least one dose of double-blind study medication and had at least one evaluable post-randomization weekly API score (i.e., where evaluable was considered a minimum of 5 diary entries in a week)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Vibegron 75 mg
Number analyzed (Participants) | 108 | 111
Participants
  IBS-D Participants: number analyzed (Participants) | 63 | 66
  IBS-D Participants | 21 | 28
  IBS-M Participants: number analyzed (Participants) | 45 | 45
  IBS-M Participants | 16 | 16
  All Participants | 37 | 44
Statistical Analysis 1: Comparison: Placebo vs Vibegron 75 mg; IBS-D Participants; Test type: Other; CMH Difference = 9.1, 90% CI 2-sided [-4.8 to 22.9] — Difference in proportion and corresponding confidence interval were calculated using the CMH risk difference estimate stratified by randomized Baseline abdominal pain (< 6 versus >= 6) strata, with weights proposed by Greenland and Robins
Statistical Analysis 2: Comparison: Placebo vs Vibegron 75 mg; IBS-M Participants; Test type: Other; CMH Difference = -0.1, 90% CI 2-sided [-16.7 to 16.4] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Vibegron 75 mg; All Participants; Test type: Other; CMH Difference = 5.3, 90% CI 2-sided [-5.4 to 15.9] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Number of IBS-D Participants Who Were API Weekly Responders With ≥ 40% Improvement Over 12 Weeks
Description: An API Weekly Responder was defined as a participant who experienced a decrease in the weekly average of "worst abdominal pain in the past 24 hours" scores of at least 40% compared with the Baseline weekly average. A participant was considered a responder over Weeks 1 to 12 if they met the criteria for at least 50% of the weeks assessed (i.e., ≥6 weeks).
Time Frame: Baseline; 12 weeks
Population: Full Analysis Set for IBS-D participants
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Vibegron 75 mg
Number analyzed (Participants) | 63 | 66
Participants | 20 | 22
Statistical Analysis 1: Comparison: Placebo vs Vibegron 75 mg; Test type: Other; CMH Difference = 1.6, 90% CI 2-sided [-11.7 to 14.9] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Number of IBS-D Participants Who Were API Weekly Responders With ≥ 50% Improvement Over 12 Weeks
Description: An API Weekly Responder was defined as a participant who experienced a decrease in the weekly average of "worst abdominal pain in the past 24 hours" scores of at least 50% compared with the Baseline weekly average. A participant was considered a responder over Weeks 1 to 12 if they met the criteria for at least 50% of the weeks assessed (i.e., ≥6 weeks).
Time Frame: Baseline; 12 weeks
Population: Full Analysis Set for IBS-D participants
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Vibegron 75 mg
Number analyzed (Participants) | 63 | 66
Participants | 13 | 18
Statistical Analysis 1: Comparison: Placebo vs Vibegron 75 mg; Test type: Other; CMH Difference = 6.7, 90% CI 2-sided [-5.5 to 18.8] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE)
Description: TEAEs are defined as events that began or worsened in severity after the first dose of the double-blind study treatment through 14 days after the last dose of study treatment.
Time Frame: from the time the participant provided informed consent to participate in the study at the Screening Visit until completion of the Safety Follow-up Call (up to Day 113 or Early Withdrawal plus 28 days)
Population: Safety Analysis Set: all participants who received at least 1 dose of study treatment. Participants were included in the treatment group corresponding to the study treatment they actually received for the analysis of safety data.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Vibegron 75 mg
Number analyzed (Participants) | 111 | 111
Participants | 37 | 37

6. Secondary Outcome: Number of Participants With Clinically Meaningful Changes From Baseline in Clinical Laboratory Values at Week 12
Description: The investigator determined whether a change was clinically meaningful.
Time Frame: Baseline; Week 12
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Vibegron 75 mg
Number analyzed (Participants) | 111 | 111
Participants | 0 | 0

7. Secondary Outcome: Number of Participants With Clinically Relevant Changes From Baseline in Vital Sign Values at Week 12
Description: Clinical relevance was determined by the investigator.
Time Frame: Baseline; Week 12
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Vibegron 75 mg
Number analyzed (Participants) | 111 | 111
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: from the time the participant provided informed consent to participate in the study at the Screening Visit until completion of the Safety Follow-up Call (up to Week 14)
Description: Treatment-emergent adverse events (TEAEs), defined as events that began or worsened in severity after the first dose of the double-blind study treatment through 14 days after the last dose of study treatment, are reported for members of the Safety Analysis Set, comprised of all participants who received at least 1 dose of study treatment. Participants were included in the treatment group corresponding to the study treatment they actually received for the analysis of safety data.
Arm/Group | Placebo | Vibegron 75 mg
All-Cause Mortality (participants affected / at risk) | 0/111 | 0/111
Serious Adverse Events (participants affected / at risk) | 1/111 | 2/111
Other Adverse Events (participants affected / at risk) | 19/111 | 13/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=111) | Vibegron 75 mg (N=111)
COVID-19 (Infections and infestations) | 0 | 1
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=111) | Vibegron 75 mg (N=111)
Constipation (Gastrointestinal disorders) | 3 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 3 | 3
Bacteriuria (Infections and infestations) | 5 | 3
Gastroenteritis (Infections and infestations) | 0 | 3
Nasopharyngitis (Infections and infestations) | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 5 | 1
Headache (Nervous system disorders) | 3 | 3
Leukocyturia (Renal and urinary disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor does not object to publication by Institution or Principal Investigator (PI) of results of the Trial based on information collected or generated by the Institution or PI. However, the Institution and PI are required to provide the Sponsor with an opportunity to review any proposed publication or other type of disclosure before it is submitted or otherwise disclosed to ensure against any inadvertent disclosure of Sponsor Confidential Information or unprotected Sponsor Inventions.

DOCUMENTS (2):
  • Study Protocol (2019-11-19): https://cdn.clinicaltrials.gov/large-docs/27/NCT03806127/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-22): https://cdn.clinicaltrials.gov/large-docs/27/NCT03806127/SAP_001.pdf